CLINICAL TRIAL: NCT01328886
Title: An Extension Study to CIGE025B1301 to Evaluate the Long-term Safety, Tolerability and Efficacy of Omalizumab in Japanese Children (6 - 15 Years) With Inadequately Controlled Allergic Asthma Despite Current Recommended Treatment
Brief Title: Long-term Safety, Tolerability and Efficacy of Omalizumab in Japanese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025B1301E1
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Asthma
Keywords: omalizumab; allergic asthma; pediatric patients
MeSH Terms: interventions — Omalizumab

ARMS (1):
- Omalizumab (Experimental)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — omalizumab lyophilized 150 mg injection

SUMMARY:
The purpose of this extension study is to assess the long-term safety and tolerability of omalizumab as an add-on therapy in Japanese pediatric patients (6 to 15 years of age) with inadequately controlled allergic asthma despite current recommended treatment by providing continued treatment with omalizumab to patients who have previously completed the core study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the core study (IGE025B1301) and who in the investigator's clinical judgment could benefit from continuous treatment of the study drug.

Exclusion Criteria:

* Patients who currently have diagnosed cancer, are currently being investigated for possible cancer or have any history of cancer.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are: women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner; women whose partners have been sterilized by vasectomy or other means; using a highly effective method of birth control; or agreeing on total abstinence and the investigator also judges that the age, career lifestyle or sexual orientation of the patient ensures compliance.
* With clinically significant uncontrolled systemic disease (eg: infection, hematological disease, renal, hepatic, coronary heart disease or other cardiovascular disease, cerebro-vascular, endocrinologic or gastrointestinal disease) after the treatment period of the core study.
* Patients with a history of major protocol violations during the core study and who are considered potentially unreliable as judged by the investigator at each site.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety and tolerability of omalizumab by measuring AEs, serious AEs, physical examination, medical history, laboratory assessments and vital signs | Every 3 months for approximately 2 years

SECONDARY OUTCOMES:
To explore the efficacy of omalizumab by JPAC questionnaire; JPAC is the Japan Pediatric Asthma Control Program (JPAC) | Every 3 months for approximately 2 years
To explore the efficacy of omalizumab by QOL questionnaire score (Quality of life questionnaires for pediatric patients with bronchial asthma and their parents or caregivers (Gifu)) | Every 3 months for approximately 2 years
To explore the efficacy of omalizumab by use of asthma long-term control medications | Every 3 months for approximately 2 years
To explore the efficacy of omalizumab by Pulmonary function (FEV1, FVC, V(・)50, V(・)25 and FEF25-75%) | Every 3 months for approximately 2 years
To collect the data on the number of hospitalizations, emergency room (ER) visits due to asthma | Every 3 months for approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Japan (14):
  - Novartis Investigative Site, Ohbu, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Shimotsuka-gun, Tochigi
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Komae, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Sumida-ku, Tokyo

REFERENCES:
- [Derived] Odajima H, Ebisawa M, Nagakura T, Fujisawa T, Akasawa A, Ito K, Doi S, Yamaguchi K, Katsunuma T, Kurihara K, Teramoto T, Sugai K, Nambu M, Hoshioka A, Yoshihara S, Sato N, Seko N, Nishima S. Long-term safety, efficacy, pharmacokinetics and pharmacodynamics of omalizumab in children with severe uncontrolled asthma. Allergol Int. 2017 Jan;66(1):106-115. doi: 10.1016/j.alit.2016.06.004. Epub 2016 Aug 6. PMID 27507228